CLINICAL TRIAL: NCT01284296
Title: Comparison of Three Methods of Hemoglobin Monitoring in Patients Undergoing Spine or Hip Surgery
Brief Title: Comparison of Three Methods of Hemoglobin Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 10-00524B
Record Dates: First submitted 2011-01-19; First posted 2011-01-26 (Estimated); Results first posted 2012-04-04 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Digital Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Digital block (Experimental)
  Interventions: Drug: Lidocaine digital block; Device: Masimo SpHb continuous hemoglobin monitor

INTERVENTIONS:
Drug: Lidocaine digital block — One dose of lidocaine 2% injected locally into one finger (2 mls total)
Device: Masimo SpHb continuous hemoglobin monitor — Masimo SpHb continuous hemoglobin monitor

SUMMARY:
This study will further investigate the Masimo SpHb [FDA Approved] continuous non-invasive hemoglobin monitor in spine surgery patients. (See NCT00792597) We will investigate the effect of enhanced circulation to the finger (which will be attached to the sensor) following a local injection (digital block) of lidocaine (an FDA approved local anesthetic), and assess the accuracy of the SpHb reading as it relates to a standard laboratory hemoglobin value (tHb).

DETAILED DESCRIPTION:
We have completed a study with 20 patients using the latest version of the SpHb monitor software and finger sensor.

The purpose of this study is to assess the accuracy of the SpHb reading as it relates to a standard laboratory hemoglobin value (tHb) following the digital block.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female 18 y/o or older
* ASA Classification 1, 2 or 3
* Scheduled to undergo spine or hip revision surgery

Exclusion Criteria:

* Pregnant or nursing
* Patients who in the study investigators clinical judgement would not be suitable for research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald D Miller, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Digital Block: The difference between intermittent readings of the SpHb continuous hemoglobin monitor with the digital lidocaine block and a laboratory hemoglobin were evaluated for patients undergoing spine surgery and blood loss.
Period: Overall Study
Arm/Group | Digital Block
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Digital Block
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Categorical Groups Based on Magnitude of Differences Between Noninvasive (SpHb) and Laboratory Co-Oximeter (tHb) Hemoglobin in Patients With a Finger Regional Anesthetic Block.
Time Frame: A minimum of 2-4 differences recorded approximately hourly during surgery
Measure: Number; unit: percentage of hemoglobin readings
Units Other Than Participants: hemoglobin readings
Groups:
- Digital Block (All Perfusion Indices 0.29-8.3): The difference between intermittent readings of the SpHb continuous hemoglobin monitor with the digital lidocaine block and a laboratory hemoglobin were evaluated for patients undergoing spine surgery and blood loss.
- Digital Block (Perfusion Indices >2.0): The difference between intermittent readings of the SpHb continuous hemoglobin monitor with the digital lidocaine block and a laboratory hemoglobin were evaluated for patients undergoing spine surgery and blood loss. This is a subgroup of differences with the perfusion index >2.0
Arm/Group | Digital Block (All Perfusion Indices 0.29-8.3) | Digital Block (Perfusion Indices >2.0)
Number analyzed (Participants) | 20 | 20
Number analyzed (hemoglobin readings) | 57 | 35
percentage of hemoglobin readings
  < 0.5 g/dL | 37 | 37
  0.5-1.0 g/dL | 19 | 26
  1.1-1.5 g/dL | 18 | 20
  1.6-2.0 g/dL | 17 | 14
  >2.0 g/dL | 9 | 3

ADVERSE EVENTS:
Arm/Group | Digital Block
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No